CLINICAL TRIAL: NCT00194246
Title: Cognitive Performance and Food Reactivity During High and Low Carbohydrate Obesity Treatment
Brief Title: Cognitive Function and Cue-Reactivity Study
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AT001103-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2007-08

CONDITIONS: Cognitive Performance; Food Cravings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — salivary cortisol
Oversight: Data Monitoring Committee: No

SUMMARY:
We are interested in testing differences in cognitive function and food reactivity at various time points in individuals following low and high carbohydrate diets. We wish to achieve an understanding of these time-specific differences using repeated measures analysis of variance (ANOVA), with diet condition (low vs. high carbohydrate) as a between subject factor and time as a within-subject factor.

DETAILED DESCRIPTION:
Participants will be recruited from the parent study The Safety and Efficacy of Low and High Carbohydrate Diets. Participants will attend one 30-minute training session to learn the computer tasks and rate food desirability. Participants will rate their desire to eat "24" foods on a "9"-point Likert scale (e.g., 1 = do not desire at all; 5 = neutral, neither desire nor not desire; 9 = desire extremely). These ratings will be used to establish emotionally salient and neutral cues for the computerized tests (i.e., Cue Reactivity and Stroop test) used during the study.

Each individual will participate on separate occasions in one 45-60 minute testing session before onset of treatment (week 0), and four 45-60 minute testing sessions that coincide with treatment assessments in the approved study (weeks 12, 26, 54). Testing will be conducted one and a half hours following consumption of a standard snack to ensure that all participants are in the same metabolic state. Participants will complete three consecutive computerized tests in the following order: 1) Continual Performance Test (CPT), 2) Stroop test, 3) Cue Reactivity Test. Based on a previous study showing impairments in cognitive function one week after initiation of a low carbohydrate diet, participants will also complete a 5-minute cognitive task (e.g., Continual Performance Task) one and four weeks after modifications in eating have begun. On these weeks, participants will be given a small snack prior to the group meeting. Testing will occur at the conclusion of weekly group meetings, ensuring that participants have abstained from food for approximately one and half hours.

The 15 minute cue reactivity test consists of three cue trials that vary only in terms of the cue presented (one neutral non-food cue, one neutral food cue, and one emotionally salient food cue). The order of these trials will be presented in a counter-balanced order.Participants will complete a VAS questionnaire, rating their feelings of hunger, craving, and anxiety. Participants will insert dental rolls prior to each of three, five-minute cue-presentation trials. While participants insert the dental rolls, the experimenter will place the relevant cue on a platter. This platter will have a divider/ barrier attached to it that obstructs the cue from the participant's view while the experimenter is in the room. After the rolls are inserted and the cue is placed on the platter, the experimenter will leave the room, and rotate the platter via remote control until the cue is in clear view of the participant.5-minute psychophysiologic data (i.e., heart rate, skin conductance) acquisition will begin as the platter is being rotated. Participants will be instructed via audiotape to focus their attention on the cue, imagine picking it up, smelling it, and tasting it, etc. At the end of this 5-minute interval, blood pressure measures will be taken.Participants will remove the dental rolls and place them in a plastic zip-lock bag.The experimenter will return to the room and ask the participant to complete the post-trial VAS questionnaire, rating their feelings of hunger, craving, and anxiety. Then participants will be provided with one ounce of water.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 30 and 40
* Live and work within 1 hour of the study site
* Stable psychological status

Exclusion Criteria:

* History of heart disease, heart attack, or stroke
* Blood pressure > 140/90 mmHG
* Abnormal cholesterol levels
* Significant psychiatric illness
* Any medication that affects weight or metabolic rate
* Presence or history of a chronic disease that is known to affect appetite, food intake, or metabolism (i.e. diabetes, thyroid disease or cancer).
* Currently using antidepressants, steroids, tobacco or illegal drugs
* Pregnant, breastfeeding, or planning pregnancy
* 10 lb change in weight within 6 months of study entry
* History of malignant arrhythmias or cerebrovascular, renal, or hepatic disease
* History of protein wasting diseases or gout
* Severe arthritis
* Osteoporosis
* Certain types of hormone replacement therapy
* Currently following a vegetarian diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all participants who took part in the Safety and Efficacy of Low and High Carbohydrate Diets study
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2003-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
the relationships between cognitive and physiological reactivity to food and non-food cues | 2 year period

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University - Center for Obesity Research and Education
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States